CLINICAL TRIAL: NCT06292520
Title: ABLLS-R and Portage Guide in the Development of Receptive Language Skills in Children With Autism Spectrum Disorder.
Brief Title: Comparison of ABLLS-R and Portage Guide in the Development of Receptive Language Skills Autism Spectrum Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4847
Record Dates: First submitted 2023-12-25; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorders; Non-verbal Learning Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABLLS-R protocol (Experimental): The study will evaluate the ABLLS-R (Assessment of Basic Language and Learning Skills test) and compare their effectiveness in developing the Receptive.
  Interventions: Other: ABLLS-R protocol
- Portage Guide Protocol (Experimental): The study will evaluate Portage guidance and compare their effectiveness in developing the Receptive Language Skills in children with Autism Spectrum Disorder.
  Interventions: Other: Portage Guide Protocol

INTERVENTIONS:
Other: Portage Guide Protocol — Portage Guide Protocol will be given to this group The study will follow the Randomized control trial study design and a purposive sampling technique will be used. Data will be collected from a special education centre BASES (Behaviour and special education services), Lahore. Children with autism spectrum disorder with mild to moderate severity level will be included in the study. The age range of the children will be from three years to seven years. Children with other neurological disorders or any comorbid conditions will be excluded from the study. The consent form will be filled out by parents of children who meet the inclusion criteria. The autism screening tool will apply by the speech and language pathologist. Half of the total number of children will receive therapeutic intervention under ABL
  Arms: Portage Guide Protocol
Other: ABLLS-R protocol — ABLLS-R protocol will be given to this group
  Arms: ABLLS-R protocol

SUMMARY:
Language is the system someone uses to communicate with another person. This covers the origins and construction of words, their definitions, and the use of language in various contexts. In normally developing children, receptive language skills are typically much more advanced than expressive language skills. However, some studies found that toddlers and kids with ASD had a relatively greater impairment in receptive language skills than in expressive language skills. The study will evaluate the ABLLS-R (Assessment of Basic Language and Learning Skills test) and Portage guidance and compare their effectiveness in developing the Receptive Language Skills in children with Autism Spectrum Disorder (N=12).

The study will follow the Randomized control trial study design and a purposive sampling technique will be used. Data will be collected from a special education centre BASES (Behaviour and special education services), Lahore. Children with autism spectrum disorder with mild to moderate severity level will be included in the study. The age range of the children will be from three years to seven years. Children with other neurological disorders or any comorbid conditions will be excluded from the study. The consent form will be filled out by parents of children who meet the inclusion criteria. The autism screening tool will apply by the speech and language pathologist. Half of the total number of children will receive therapeutic intervention under ABLLS-R protocol and other will receive Interventions under portage guide protocol. The data will be analysed by using SPSS 22 statistical software. The results of the study of both the groups will be compared and conclusion will be made on the basis of results. Receptive language skills are crucial for communication and social interaction. Research comparing these assessment tools can contribute to the development of more effective early intervention programs for children with ASD. By identifying the most appropriate assessment tool and intervention strategies, these programs can be better designed to support early language development and promote better long-term outcomes. By understanding the strengths and limitations of each assessment tool, professionals can create more individualized treatment plans for children with ASD

ELIGIBILITY:
Inclusion Criteria:

* Children with autism spectrum disorder with mild to moderate severity level will be included in the study.
* The age range of the children will be from three years to seven years.

Exclusion Criteria:

* Children with other neurological disorders or any comorbid conditions will be excluded from the study.
* Children who are not participated in any kind of other intervention.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
ABLLS-R for the development of receptive language in children with Autism | 6 months
  Assessment of Basic Language and Learning Skills-Revised (ABLLS-R) is a criterion referenced assessment tool, curriculum planning manual, and tracking system for the prerequisite skills required for the development of basic language and communication as well as skills required to support learning in significant academic, adaptive, and motor domains assessment tool and intervention strategies, these programs can be better designed to support early language development and promote better long-term outcomes.
Portage Guide for the development of receptive language in children with Autism | 6 months
  A home-based early intervention program called Portage Guide to Early Education is for preschoolers who are developmentally delayed. It consists of a method of teaching parents how to instruct their own children, a set of reading materials, and the triadic model of service delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Aleena Irum, MS-SLP, Principal Investigator — Riphah International University
Locations (1):
- Bases Institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maljaars J, Noens I, Scholte E, van Berckelaer-Onnes I. Language in low-functioning children with autistic disorder: differences between receptive and expressive skills and concurrent predictors of language. J Autism Dev Disord. 2012 Oct;42(10):2181-91. doi: 10.1007/s10803-012-1476-1. PMID 22350453
- [Background] Sket GM, Overfeld J, Styner M, Gilmore JH, Entringer S, Wadhwa PD, Rasmussen JM, Buss C. Neonatal White Matter Maturation Is Associated With Infant Language Development. Front Hum Neurosci. 2019 Dec 17;13:434. doi: 10.3389/fnhum.2019.00434. eCollection 2019. PMID 31920593
- [Background] Plesa Skwerer D, Jordan SE, Brukilacchio BH, Tager-Flusberg H. Comparing methods for assessing receptive language skills in minimally verbal children and adolescents with autism spectrum disorders. Autism. 2016 Jul;20(5):591-604. doi: 10.1177/1362361315600146. Epub 2015 Sep 25. PMID 26408635
- [Background] Lord C, Elsabbagh M, Baird G, Veenstra-Vanderweele J. Autism spectrum disorder. Lancet. 2018 Aug 11;392(10146):508-520. doi: 10.1016/S0140-6736(18)31129-2. Epub 2018 Aug 2. PMID 30078460